CLINICAL TRIAL: NCT00577161
Title: Fludarabine, BBR 2778 (Pixantrone) and Rituximab (FP-R) vs Fludarabine and Rituximab (F-R) for Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Brief Title: Fludarabine, Pixantrone and Rituximab vs Fludarabine and Rituximab forRelapsed or Refractory Indolent NHL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: closed to enrollment
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIX303
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: pixantrone; NHL; rituximab; fludarabine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine; Rituximab; pixantrone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comparator (Active Comparator): fludarabine and rituximab
  Interventions: Drug: fludarabine and rituximab
- Experimental (Experimental): fludarabine, rituximab, pixantrone
  Interventions: Drug: fludarabine, rituximab, pixantrone

INTERVENTIONS:
Drug: fludarabine and rituximab — days 1 to 4 of six 28-day cycles rituximab 375 mg/m2 fludarabine 25 mg/m2
  Arms: Comparator
Drug: fludarabine, rituximab, pixantrone — days 1 to 4 of six 28-day cycles rituximab 375 mg/m2 fludarabine 25 mg/m2 pixantrone 120 mg/m2 day 2 only
  Arms: Experimental

SUMMARY:
BBR 2778 is a novel aza-anthracenedione that has activity in experimental tumors and reduced delayed cardiotoxicity in animal models compared to reference standards. This cytotoxic agent has structural similarities to mitoxantrone as well as general similarities to anthracyclines (such as the tricyclic central quinoid chromophore7).

This phase III study will compare the efficacy and safety of the combination BBR 2778, fludarabine, and rituximab with the combination fludarabine and rituximab in patients with relapsed or refractory indolent non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed relapsed or refractory indolent non-Hodgkin's lymphoma (NHL)
2. Any stage (Ann Arbor staging, Appendix 15.7), with or without B symptoms
3. CD 20+ lymphoma (confirmed by immunochemistry)
4. Measurable disease.
5. Atleast 1 prior therapy.
6. Age ≥ 18 years
7. Life expectancy of at least 3 months
8. ECOG performance status (PS) of 0 or 1
9. Adequate cardiac function defined as LVEF ≥ 50% by MUGA scan
10. Adequate renal function
11. Adequate hepatic function
12. Adequate bone marrow function
13. Recovery from all acute toxicities from prior therapies (except alopecia and grade 1 peripheral neuropathy).

Exclusion Criteria

1. Prior treatment with a cumulative dose of doxorubicin equivalent exceeding 450 mg/m2
2. Radiotherapy, chemotherapy or other therapies for NHL within 4 weeks of treatment start
3. Systemic corticosteroids to treat NHL within 5 days prior to first dose of study treatment.
4. Radioimmunotherapy (RIT) within 3 months of treatment start
5. Known hypersensitivity to the excipients or the study drugs that the patient will receive
6. Known Type I hypersensitivity or anaphylactic reactions to murine proteins or to any component of rituximab
7. Major thoracic and/or abdominal surgery in the preceding 4 weeks, from which the patient has not fully recovered (patients who have had minor surgery and one week's recovery period may be enrolled)
8. HIV-related lymphoma
9. Active CNS involvement
10. Clinically significant cardiovascular abnormalities
11. Serious (NCI CTCAE grade 3-4) intercurrent infection at randomization, infection requiring oral antibiotics, or deep-seated or systemic mycotic infections.
12. Investigational study drug within 30 days before randomization. Patient must have recovered from all side effects of other investigational therapy.
13. Clinical symptoms suggesting unresolved HIV, HBV or HCV infection. .
14. History of another malignancy except: curatively treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in remission, or any other cancer from which the patient has been disease-free for 5 years
15. Pregnant or lactating women
16. Potentially fertile men and women and their sexual partners not willing to use adequate contraception as defined by the Investigator during the study and for 6 months after the last day of study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
progression-free survival | day 64-71

SECONDARY OUTCOMES:
response rate, survival, safety | every 21 days

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Ventura County Hematology Oncology Specialist, Oxnard, California
  - Capitol Comprehensive Cancer Care, Jefferson City, Missouri
  - Heartland Hematology Oncology Associates, Kansas City, Missouri
  - Cancer Care Center, Albany, New York
  - Interlakes Foundation, Inc., Rochester, New York
  - Hematology Oncology Consultants, Columbus, Ohio
  - Utah Hematology Oncology, P.C., Ogden, Utah